CLINICAL TRIAL: NCT06656650
Title: Commensality Groups: A Professional Fulfillment Intervention for Medical Students in Their Clinical Years
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Chantal Sheridan, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-24-00919
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Professional Fulfillment; Burnout; Social Isolation or Loneliness
Keywords: commensality groups; medical students
MeSH Terms: conditions — Burnout, Psychological; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Participants attend commensality groups
  Interventions: Behavioral: Commensality groups
- Waitlist control group (No Intervention): Participants receive no intervention

INTERVENTIONS:
Behavioral: Commensality groups — Participants will attend at least 3 out of 6 commensality groups over the course of 6 months.
  Arms: Treatment group

SUMMARY:
Medical students are at high risk for burnout, depression, anxiety, suicidal ideation and substance use disorder with burnout seen as a mitigating factor for suicidal ideation. Help-seeking among medical students suffering from burnout is only 30%. The highest rates of burnout among medical students is at the end of their clinical rotations, with estimates of up to 60%. "Commensality groups" have been found to significantly reduce burnout and improve meaning in work by creating opportunity for connection and collegiality among physicians. These groups consist of providing a reimbursed monthly meal with structured questions that generate conversation for the first 15 minutes with 6-8 participants meeting monthly, for six months. Physician participants in Commensality groups maintain these gains one year later.

The investigators propose to apply the model of Commensality groups to medical students who are launching into their experience clinical practice, and have been on clinical rotations for at least 4 months. The investigators will form randomly assigned groups of 6-8 medical students with 1 resident leader. The resident leader role has been added to encourage compliance with the standardized discussion questions and to avoid the potential negative impact of a "venting" session. The overall intention of this study is to explore whether Commensality groups can increase well-being for medical students in their clerkship years, as it has previously been shown to do for residents and physicians.

ELIGIBILITY:
Inclusion Criteria:

* Currently a medical student on clerkships at the Keck School of Medicine of the University of Southern California

Exclusion Criteria:

* Not currently on a leave of absence, research year, or otherwise not enrolled in the medical school program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Survey | Baseline (within one month prior to launch of study), immediately post intervention (within one month after final intervention), approximately 3 months after the final intervention, and approximately 6 months after the final intervention
  Survey containing 5 evidence-based measures

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Sheridan, PhD, Principal Investigator — Keck School of Medicine, University of Southern California; Maria Juliani, PhD, Study Director — Keck School of Medicine, University of Southern California
Locations (1):
- Keck School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for all study participants will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Hansell MW, Ungerleider RM, Brooks CA, Knudson MP, Kirk JK, Ungerleider JD. Temporal Trends in Medical Student Burnout. Fam Med. 2019 May;51(5):399-404. doi: 10.22454/FamMed.2019.270753. PMID 31081911
- [Background] Dyrbye L, Shanafelt T. A narrative review on burnout experienced by medical students and residents. Med Educ. 2016 Jan;50(1):132-49. doi: 10.1111/medu.12927. PMID 26695473
- [Background] Dyrbye LN, Thomas MR, Massie FS, Power DV, Eacker A, Harper W, Durning S, Moutier C, Szydlo DW, Novotny PJ, Sloan JA, Shanafelt TD. Burnout and suicidal ideation among U.S. medical students. Ann Intern Med. 2008 Sep 2;149(5):334-41. doi: 10.7326/0003-4819-149-5-200809020-00008. PMID 18765703
- [Background] Dyrbye LN, Thomas MR, Shanafelt TD. Systematic review of depression, anxiety, and other indicators of psychological distress among U.S. and Canadian medical students. Acad Med. 2006 Apr;81(4):354-73. doi: 10.1097/00001888-200604000-00009. PMID 16565188
- [Background] Rotenstein LS, Ramos MA, Torre M, Segal JB, Peluso MJ, Guille C, Sen S, Mata DA. Prevalence of Depression, Depressive Symptoms, and Suicidal Ideation Among Medical Students: A Systematic Review and Meta-Analysis. JAMA. 2016 Dec 6;316(21):2214-2236. doi: 10.1001/jama.2016.17324. PMID 27923088
- [Background] Dyrbye LN, Eacker A, Durning SJ, Brazeau C, Moutier C, Massie FS, Satele D, Sloan JA, Shanafelt TD. The Impact of Stigma and Personal Experiences on the Help-Seeking Behaviors of Medical Students With Burnout. Acad Med. 2015 Jul;90(7):961-9. doi: 10.1097/ACM.0000000000000655. PMID 25650824
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053